CLINICAL TRIAL: NCT03031093
Title: Aerosol Therapy With High Flow Nasal Cannula (HFNC) in Obese COPD Patients. Aerosol Deposition Pattern and Predictive Values.
Brief Title: Aerosol Therapy in Obese COPD Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Taciano Dias de Souza Rocha, Master in Physiotherapy, Universidade Federal do Rio Grande do Norte
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: CAAE: 57946516.0.0000.5537
Record Dates: First submitted 2016-12-06; First posted 2017-01-25 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Chronic Obstructive Pulmonary Disease Moderate; Obesity
Keywords: aerosol therapy; pulmonary scintigraphy; upper airways anatomy; High Flow Nasal Cannula
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Healthy, non obese + HFNC (Experimental): Healthy, non obese participants will perform the following inhalation protocol:aerosol solution of technetium labeled diethylenetriaminepenta-acetic acid (99mTc-DTPA) (1mCi) and bronchodilators (fenoterol (2.5 mg) and ipratropium bromide (0.25 mg)) with 0.9% saline solution (total 1,5 ml) using a vibrating MESH inhaler (Aerogen® Solo, Aerogen Ltd, Galway, Ireland). A High Flow Nasal Cannula (HFNC) with 30L/min flow will be used to deliver aerosol. Volunteer seated; Preliminary acclimatization (1-2 min). Inspiratory branch: source of oxygen; HFNC; Expiratory branch: filter (Vital signs, USA). Nebulization will run until the full dose has been used (3-4 min).
  Interventions: Radiation: inhalation protocol; Device: High Flow Nasal Cannula
- Healthy, non obese (Active Comparator): Healthy, non obese participants will perform the following inhalation protocol: aerosol solution of technetium labeled diethylenetriaminepenta-acetic acid (99mTc-DTPA) (1mCi) and bronchodilators (fenoterol (2.5 mg) and ipratropium bromide (0.25 mg)) with 0.9% saline solution (total dose volume 1,5 ml) using a vibrating MESH inhaler (Aerogen® Solo, Aerogen Ltd, Galway, Ireland) with free flow. The volunteer will be positioned seated in a chair. A mouthpiece associated with a T-tube with Inspiratory and Expiratory branches will be positioned in his mouth for preliminary acclimatization (1-2 min). Inspiratory branch: source of oxygen; bag of air accumulation. Expiratory branch: filter (Vital signs, USA). Nebulization will run until the full dose has been used (3-4 min).
  Interventions: Radiation: inhalation protocol
- COPD, non obese + HFNC (Experimental): non obese COPD participants will perform the following inhalation protocol:aerosol solution of technetium labeled diethylenetriaminepenta-acetic acid (99mTc-DTPA) (1mCi) and bronchodilators (fenoterol (2.5 mg) and ipratropium bromide (0.25 mg)) with 0.9% saline solution (total 1,5 ml) using a vibrating MESH inhaler (Aerogen® Solo, Aerogen Ltd, Galway, Ireland). A High Flow Nasal Cannula (HFNC) with 30L/min flow will be used to deliver aerosol. Volunteer seated; Preliminary acclimatization (1-2 min). Inspiratory branch: source of oxygen; HFNC; Expiratory branch: filter (Vital signs, USA). Nebulization will run until the full dose has been used (3-4 min).
  Interventions: Radiation: inhalation protocol; Device: High Flow Nasal Cannula
- COPD, non obese (Active Comparator): non obese COPD participants will perform the following inhalation protocol: aerosol solution of technetium labeled diethylenetriaminepenta-acetic acid (99mTc-DTPA) (1mCi) and bronchodilators (fenoterol (2.5 mg) and ipratropium bromide (0.25 mg)) with 0.9% saline solution (total dose volume 1,5 ml) using a vibrating MESH inhaler (Aerogen® Solo, Aerogen Ltd, Galway, Ireland) with free flow. The volunteer will be positioned seated in a chair. A mouthpiece associated with a T-tube with Inspiratory and Expiratory branches will be positioned in his mouth for preliminary acclimatization (1-2 min). Inspiratory branch: source of oxygen; bag of air accumulation. Expiratory branch: filter (Vital signs, USA). Nebulization will run until the full dose has been used (3-4 min).
  Interventions: Radiation: inhalation protocol
- healthy, obese + HFNC (Experimental): Healthy obese participants will perform the following inhalation protocol:aerosol solution of technetium labeled diethylenetriaminepenta-acetic acid (99mTc-DTPA) (1mCi) and bronchodilators (fenoterol (2.5 mg) and ipratropium bromide (0.25 mg)) with 0.9% saline solution (total 1,5 ml) using a vibrating MESH inhaler (Aerogen® Solo, Aerogen Ltd, Galway, Ireland). A High Flow Nasal Cannula (HFNC) with 30L/min flow will be used to deliver aerosol. Volunteer seated; Preliminary acclimatization (1-2 min). Inspiratory branch: source of oxygen; HFNC; Expiratory branch: filter (Vital signs, USA). Nebulization will run until the full dose has been used (3-4 min).
  Interventions: Radiation: inhalation protocol; Device: High Flow Nasal Cannula
- healthy, obese (Active Comparator): Healthy obese participants will perform the following inhalation protocol: aerosol solution of technetium labeled diethylenetriaminepenta-acetic acid (99mTc-DTPA) (1mCi) and bronchodilators (fenoterol (2.5 mg) and ipratropium bromide (0.25 mg)) with 0.9% saline solution (total dose volume 1,5 ml) using a vibrating MESH inhaler (Aerogen® Solo, Aerogen Ltd, Galway, Ireland) with free flow. The volunteer will be positioned seated in a chair. A mouthpiece associated with a T-tube with Inspiratory and Expiratory branches will be positioned in his mouth for preliminary acclimatization (1-2 min). Inspiratory branch: source of oxygen; bag of air accumulation. Expiratory branch: filter (Vital signs, USA). Nebulization will run until the full dose has been used (3-4 min).
  Interventions: Radiation: inhalation protocol
- COPD, obese + HFNC (Experimental): Obese COPD participants will perform the following inhalation protocol:aerosol solution of technetium labeled diethylenetriaminepenta-acetic acid (99mTc-DTPA) (1mCi) and bronchodilators (fenoterol (2.5 mg) and ipratropium bromide (0.25 mg)) with 0.9% saline solution (total 1,5 ml) using a vibrating MESH inhaler (Aerogen® Solo, Aerogen Ltd, Galway, Ireland). A High Flow Nasal Cannula (HFNC) with 30L/min flow will be used to deliver aerosol. Volunteer seated; Preliminary acclimatization (1-2 min). Inspiratory branch: source of oxygen; HFNC; Expiratory branch: filter (Vital signs, USA). Nebulization will run until the full dose has been used (3-4 min).
  Interventions: Radiation: inhalation protocol; Device: High Flow Nasal Cannula
- COPD, obese (Active Comparator): Obese COPD participants will perform the following inhalation protocol:aerosol solution of technetium labeled diethylenetriaminepenta-acetic acid (99mTc-DTPA) (1mCi) and bronchodilators (fenoterol (2.5 mg) and ipratropium bromide (0.25 mg)) with 0.9% saline solution (total 1,5 ml) using a vibrating MESH inhaler (Aerogen® Solo, Aerogen Ltd, Galway, Ireland). The volunteer will be positioned seated in a chair. A mouthpiece associated with a T-tube with Inspiratory and Expiratory branches will be positioned in his mouth for preliminary acclimatization (1-2 min). Inspiratory branch: source of oxygen; bag of air accumulation. Expiratory branch: filter (Vital signs, USA). Nebulization will run until the full dose has been used (3-4 min).
  Interventions: Radiation: inhalation protocol

INTERVENTIONS:
Radiation: inhalation protocol — technetium labeled diethylenetriaminepenta-acetic acid (99mTc-DTPA) (1mCi) and bronchodilators (fenoterol (2.5 mg) and ipratropium bromide (0.25 mg)) with 0.9% saline solution
Device: High Flow Nasal Cannula — aerosol solution of technetium labeled diethylenetriaminepenta-acetic acid (99mTc-DTPA) (1mCi) and bronchodilators (fenoterol (2.5 mg) and ipratropium bromide (0.25 mg)) with 0.9% saline solution (total 1,5 ml) using a vibrating MESH inhaler (Aerogen® Solo, Aerogen Ltd, Galway, Ireland). A High Flow Nasal Cannula will deliver the aerosol at a 30L/min flow of oxigen.
  Arms: COPD, non obese + HFNC; COPD, obese + HFNC; Healthy, non obese + HFNC; healthy, obese + HFNC

SUMMARY:
This study has the objective to clarify the factors that directly influence the effectiveness of inhaled drug deposition in obese patients with chronic obstructive pulmonary disease (COPD) and suggest the use of High Flow Nasal Cannula (HFNC) during their inhalation therapy.

DETAILED DESCRIPTION:
This study has the objective to clarify the factors that directly influence the effectiveness of inhaled drug deposition in obese patients with chronic obstructive pulmonary disease (COPD) and then formulate specific strategies to control the evolution of this disease. The suggested strategy in order to implement the aerosol therapy is the use of High Flow Nasal Cannula (HFNC) during these patient´s inhalation therapy.

It will consist in a cross-over clinical trial. The population will be composed by volunteers of both genders, aged between 45-70 years old. Four distinct groups will be formed: obese participants without copd; obese participants with copd; non obese participants without copd; non-obese participants with copd.

ELIGIBILITY:
Inclusion Criteria:

HEALTHY, non obese

* no history of respiratory disease
* non smokers
* self declared sedentary
* Forced expiratory volume at first second (FEV1) equal or higher than 80% of predicted
* Forced Vital capacity (FVC) equal or higher than 80% of predicted;
* FEV1/FVC higher than 70% of predicted.
* BMI lower than 30 kg/m2

HEALTHY, obese

* no history of respiratory disease
* non smokers
* self declared sedentary
* Forced expiratory volume at first second (FEV1) equal or higher than 80% of predicted
* Forced Vital capacity (FVC) equal or higher than 80% of predicted
* FEV1/FVC higher than 70% of predicted.
* BMI equal or higher than 30 kg/m2

COPD participants, non obese

* ex smokers
* clinical stability (six previous weeks)
* FEV1 lower than 80% of predicted.
* FEV1/FVC lower than 70 % post bronchodilator.
* No cardiopulmonary diseases (self declared)
* BMI lower than 30 kg/m2

COPD participants, obese

* ex smokers
* clinical stability (six previous weeks)
* FEV1 lower than 80% of predicted.
* FEV1/FVC lower than 70 % post bronchodilator.
* No cardiopulmonary diseases (self declared)
* BMI equal or higher than 30 kg/m2

Exclusion Criteria:

* Difficulty to understand verbal commands
* exacerbations during the study period

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-12-02 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2018-05-05 (Actual)

PRIMARY OUTCOMES:
Pattern of aerosol lung deposition. | during the following 25 minutes post inhalation protocol
  The pattern of aerosol lung deposition will be compared between obese and non obese participants (with and without COPD) as well as between inhalation with HFNC and without HFNC

SECONDARY OUTCOMES:
Change of pulmonary function after bronchodilators administration. (with and without HFNC) | Change from Baseline Pulmonary Function at 5 minutes after scintigraphy.
  pulmonary function will be evaluated previously to the inhalation protocol. After the inhalation protocol, this measurement will be assessed again in order to check the effect of bronchodilator drug.
Upper airways anatomical variables CT scans | first day of study
  Upper airways anatomical variables will be measured by CT scans.
Mallampati Score | first day of study
  Mallampati Score (from 1 to 4)
BMI | first day of study
  Body mass index
Muscle Mass | first day of study
  Muscle Mass percentage
Body fat | first day of study
  Body fat percentage

CONTACTS AND LOCATIONS:
Overall Officials: Armele Dornelas de Andrade, PhD, Study Director — Universidade Federal de Pernambuco
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rocha T, Rattes C, Morais C, Souza R, Rolim N, Brandao S, Fink JB, Dornelas de Andrade A. Predictive anatomical factors of lung aerosol deposition in obese individuals. Would modified mallampati score be relevant? Clinical trial. Respir Med. 2020 Sep;171:106083. doi: 10.1016/j.rmed.2020.106083. Epub 2020 Jul 12. PMID 32917355